CLINICAL TRIAL: NCT05899829
Title: A Phase 1, 2-part, Open-label, Fixed-sequence Study Evaluating the Effect of Rifampin (Part 1) and Rabeprazole (Part 2) on the Pharmacokinetics of a Single Dose of Camlipixant (BLU-5937) 50 mg Tablet in Healthy Participants Under Fasting Conditions
Brief Title: Evaluation of the Effect of Rifampin and Rabeprazole on the Pharmacokinetics of Camlipixant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221853; BUS-P1-11 (Other: Bellus Health Inc)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Cough; Healthy
MeSH Terms: conditions — Cough | interventions — Rabeprazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Camlipixant 50 mg + Rifampin 600 mg (Experimental): Participants will receive a single oral dose of camlipixant 50 milligram (mg) tablet on Day 1, followed by repeat oral doses (2*300 mg) of rifampin 600 mg capsules, once daily (QD) from Days 4 to 12, with co-administration of a single oral dose of 50 mg camlipixant tablet with rifampin capsules on Day 11. There will be a washout of at least 3 days between the dose of camlipixant on Day 1 and the dose of rifampin on Day 4.
  Interventions: Drug: Camlipixant; Drug: Rifampin
- Part 2: Camlipixant 50 mg + Rabeprazole 20 mg (Experimental): Participants will receive a single oral dose of camlipixant 50 mg tablet on Day 1, followed by repeat oral doses of 20 mg rabeprazole enteric-coated tablets, once daily (QD) from Days 4 to 11, with co-administration of a single oral dose of 50 mg camlipixant tablet with rabeprazole enteric-coated tablet on Day 10. There will be a washout of at least 3 days between the dose of camlipixant on Day 1 and the dose of rabeprazole on Day 4
  Interventions: Drug: Camlipixant; Drug: Rabeprazole

INTERVENTIONS:
Drug: Camlipixant — Camlipixant will be administered
Drug: Rabeprazole — Rabeprazole will be administered
  Arms: Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Drug: Rifampin — Rifampin will be administered.
  Arms: Part 1: Camlipixant 50 mg + Rifampin 600 mg

SUMMARY:
This is a phase 1, 2-part, open-label, fixed-sequence study evaluating the effect of rifampin (part 1) and rabeprazole (part 2) on the pharmacokinetics of a single dose of camlipixant (BLU-5937) 50 mg tablet in healthy participants under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females

Exclusion Criteria:

* History of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disorder, as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 42 participants were enrolled (20 participants in Part 1 and 22 participants in Part 2) in this study. Only 32 participants (10 participants were never dosed) were dosed into the study to receive either camlipixant + rifampin or camlipixant + rabeprazole creating the Safety Population.
Groups:
- Part 1: Camlipixant 50 mg + Rifampin 600 mg: Participants received a single oral dose of camlipixant 50 milligram (mg) tablet on Day 1, followed by repeat oral doses (2*300 mg) of rifampin 600 mg capsules, once daily (QD) from Days 4 to 12, with co-administration of a single oral dose of 50 mg camlipixant tablet with rifampin capsules on Day 11. There was a washout of at least 3 days between the dose of camlipixant on Day 1 and the dose of rifampin on Day 4.
- Part 2: Camlipixant 50 mg + Rabeprazole 20 mg: Participants received a single oral dose of camlipixant 50 mg tablet on Day 1, followed by repeat oral doses of 20 mg rabeprazole enteric-coated tablets, once daily (QD) from Days 4 to 11, with co-administration of a single oral dose of 50 mg camlipixant tablet with rabeprazole enteric-coated tablet on Day 10. There was a washout of at least 3 days between the dose of camlipixant on Day 1 and the dose of rabeprazole on Day 4.
Period: Part 1 (Up to Day 22)
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Started (Enrolled) | 20 | 0
Safety Population | 16 | 0
Completed | 16 | 0
Not Completed | 4 | 0
Not completed — Enrolled but did not receive study treatment | 4 | 0
Period: Part 2 (up to Day 21)
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Started (Enrolled) | 0 | 22
Safety Population | 0 | 16
Completed | 0 | 16
Not Completed | 0 | 6
Not completed — Enrolled but did not receive study treatment | 0 | 6

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the Safety Population which consisted of all participants who received at least one dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Customized [Count of Participants; unit: Participants]
  18 to 55 years | 16 | 16 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 15 | 11 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories (with 0<n<11) are combined into 'Others' category to maintain participant confidentiality and privacy.
  Participants
    Others | 1 | 1 | 2
    White | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC[0-Infinity]) of Camlipixant
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of Camlipixant. PK analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 0.16, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 36, and 48 hours post-dose on Day 1 and Day 11
Population: Pharmacokinetic Parameter Population comprised of all participants for whom the Day 1 and Day 11 (Part 1) PK profiles of Camlipixant were adequately characterized, specifically, when administered alone and in combination with Rifampin (Part 1).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Hours*nanograms per milliliter
  Day 1 | 3851.24 (39.27)
  Day 11 | 1423.84 (38.90)

2. Primary Outcome: Part 2: AUC(0-Infinity) of Camlipixant
Description: Blood samples were collected at indicated time points for PK analysis of Camlipixant. PK analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 0.16, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15, 18, 24, 36, and 48 hours post-dose on Day 1 and Day 10
Population: Pharmacokinetic Parameter Population comprised of all participants for whom the Day 1 and Day 10 (Part 2) PK profiles of Camlipixant, were adequately characterized, specifically, when administered alone and in combination with Rabeprazole (Part 2).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Hours*nanograms per milliliter
  Day 1 | 5425.54 (29.55)
  Day 10 | 5514.74 (33.39)

3. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero Until the Last Observed Concentration (AUC[0-t]) of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Hours*nanograms per milliliter
  Day 1 | 3834.41 (39.31)
  Day 11 | 1419.39 (38.97)

4. Primary Outcome: Part 2: AUC(0-t) of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Hours*nanograms per milliliter
  Day 1 | 5403.91 (29.52)
  Day 10 | 5474.24 (33.07)

5. Primary Outcome: Part 1: Maximum Observed Concentration (Cmax) of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Nanograms per milliliter
  Day 1 | 819 (19.54)
  Day 11 | 519 (27.84)

6. Primary Outcome: Part 2: Cmax of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Nanograms per milliliter
  Day 1 | 1080 (24.74)
  Day 10 | 912 (34.29)

7. Secondary Outcome: Part 1: Time to Reach Maximum Observed Concentration (Tmax) of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Hours
  Day 1 | 1.000 [0.250 to 2.500]
  Day 11 | 0.750 [0.500 to 3.000]

8. Secondary Outcome: Part 2: Tmax of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Hours
  Day 1 | 0.750 [0.500 to 1.000]
  Day 10 | 1.750 [0.600 to 4.017]

9. Secondary Outcome: Part 1: Terminal Elimination Half-Life (T1/2) Following Administration of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Hours
  Day 1 | 5.05 (32.02)
  Day 11 | 1.94 (28.68)

10. Secondary Outcome: Part 2: T1/2 Following Administration of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Hours
  Day 1 | 6.01 (16.90)
  Day 10 | 6.78 (17.01)

11. Secondary Outcome: Part 1: Percentage of AUC0-Infinity Due to Extrapolation From the Time of the Last Observed Concentration to Infinity (% AUC Extrapolation) of Camlipixant
Description: Blood samples were collected at indicated time points for PK analysis of Camlipixant. PK analysis was conducted using standard non-compartmental methods. Percentage of AUC extrapolation was calculated as [1 - (AUC0-t/AUC0-inf)] * 100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolation
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Percentage of AUC extrapolation
  Day 1 | 0.40 (45.60)
  Day 11 | 0.30 (33.74)

12. Secondary Outcome: Part 2: % AUC Extrapolation of Camlipixant
Description: as for outcome 11
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolation
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Percentage of AUC extrapolation
  Day 1 | 0.34 (54.00)
  Day 10 | 0.57 (84.03)

13. Secondary Outcome: Part 1: Terminal Elimination Rate Constant of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Per hour
  Day 1 | 0.1372 (32.02)
  Day 11 | 0.3579 (28.68)

14. Secondary Outcome: Part 2: Terminal Elimination Rate Constant of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Per hour
  Day 1 | 0.1153 (16.90)
  Day 10 | 0.1022 (17.01)

15. Secondary Outcome: Part 1: Apparent Clearance (CL/F) of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Liters per hour
  Day 1 | 12.98 (39.27)
  Day 11 | 35.12 (38.90)

16. Secondary Outcome: Part 2: CL/F of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Liters per hour
  Day 1 | 9.22 (29.55)
  Day 10 | 9.07 (33.39)

17. Secondary Outcome: Part 1: Apparent Oral Volume of Distribution (Vz/F) of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Liters
  Day 1 | 94.66 (26.40)
  Day 11 | 98.11 (29.90)

18. Secondary Outcome: Part 2: Vz/F of Camlipixant
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Liters
  Day 1 | 79.96 (31.72)
  Day 10 | 88.74 (26.78)

19. Secondary Outcome: Part 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs) and Treatment-emergent Adverse Events of Medical Interest (TEAEMIs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant who is administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. Serious adverse events (SAEs) are defined as any untoward medical occurrence that; at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. Adverse events of medical interest (AEMIs) are AEs of scientific interest specific to the drug class. Treatment-emergent events (i.e., TEAEs, TESAEs and TEAEMIs) were defined as events that commence on or after the time of first study drug administration.
Time Frame: Up to Day 22 for Part1 (Day1 post-dose until Day4 pre-dose of rifampin [Camlipixant 50mg];From Day4 dosing until Day11 pre-dose of camlipixant [Rifampin 600mg];From camlipixant dosing on Day11 until end of study [Day 22] [Camlipixant 50mg+Rifampin 600mg]
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Camlipixant 50 mg: Participants received a single oral dose of 50 mg camlipixant tablet on Day 1.
- Part 1: Rifampin 600 mg: Participants received repeated oral doses of 2*300 mg rifampin capsules (total dose 600 mg) once daily on Days 4 to 12.
- Part 1: Camlipixant 50 mg+ Rifampin 600 mg: Participants received repeat oral doses (2*300 mg) of rifampin 600 mg capsules, once daily (QD) from Days 4 to 12, with co-administration of a single oral dose of 50 mg camlipixant tablet with rifampin capsules on Day 11.Participants were followed up for adverse events until end of study (up to Day 22)
Arm/Group | Part 1: Camlipixant 50 mg | Part 1: Rifampin 600 mg | Part 1: Camlipixant 50 mg+ Rifampin 600 mg
Number analyzed (Participants) | 16 | 16 | 16
Participants
  TEAEs | 3 | 14 | 2
  TESAEs | 0 | 0 | 0
  TEAEMIs | 0 | 0 | 0

20. Secondary Outcome: Part 2: Number of Participants With TEAEs, TESAEs and TEAEMIs
Description: as for outcome 19
Time Frame: Upto Day21 for Part2(Day1 postdose until Day4 predose of rabeprazole [Camlipixant 50mg];From Day4 dosing until Day10 predose of camlipixant [Rabeprazole 20mg];From camlipixant dosing on Day10 until end of study[Day21] [Camlipixant 50mg+Rabeprazole 20mg]
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Camlipixant 50 mg: Participants received a single oral dose of 50 mg camlipixant tablet on Day 1.
- Part 2 : Rabeprazole 20 mg: Participants received repeated oral doses of 1*20 mg rabeprazole enteric-coated tablets once daily on Days 4 to 11.
- Part 2: Camlipixant 50 mg+ Rabeprazole 20 mg: Participants received repeat oral doses of 20 mg rabeprazole enteric-coated tablets, once daily (QD) from Days 4 to 11, with co-administration of a single oral dose of 50 mg camlipixant tablet with rabeprazole enteric-coated tablet on Day 10. Participants were followed up for adverse events until end of study (up to Day 21)
Arm/Group | Part 2: Camlipixant 50 mg | Part 2 : Rabeprazole 20 mg | Part 2: Camlipixant 50 mg+ Rabeprazole 20 mg
Number analyzed (Participants) | 16 | 16 | 16
Participants
  TEAEs | 4 | 3 | 0
  TESAEs | 0 | 0 | 0
  TEAEMIs | 0 | 0 | 0

21. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in 12-Lead Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded with the participant in a semi-recumbent or supine position, after 5 minutes of rest using an ECG machine. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant 12-Lead ECG findings have been presented.
Time Frame: Day 4, Day 11, and Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Participants
  Day 4 | 0
  Day 11 | 0
  Day 13 | 0

22. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in 12-Lead ECG Findings
Description: as for outcome 21
Time Frame: Day 4, Day 10, and Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Participants
  Day 4 | 0
  Day 10 | 0
  Day 12 | 0

23. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Vital Signs: Diastolic Blood Pressure (DBP), Systolic Blood Pressure (SBP), and Heart Rate
Description: Vital signs including diastolic blood pressure (DBP), systolic Blood Pressure (SBP), and heart rate were measured in a sitting position after resting for at least 5 minutes. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant changes for vital signs have been presented.
Time Frame: Day 11 and Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Participants
  Day 11 | 0
  Day 13 | 0

24. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Vital Signs: DBP, SBP, and Heart Rate
Description: Vital signs including DBP, SBP, and heart rate were measured in a sitting position after resting for at least 5 minutes. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant changes for vital signs have been presented.
Time Frame: Day 10 and Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Participants
  Day 10 | 0
  Day 12 | 0

25. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Vital Signs: Respiratory Rate and Oral Temperature
Description: Vital signs including respiratory rate and oral temperature were measured after resting for at least 5 minutes in a sitting position. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant changes for vital signs have been presented.
Time Frame: Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Participants | 0

26. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Vital Signs: Respiratory Rate and Oral Temperature
Description: as for outcome 25
Time Frame: Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Participants | 0

27. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Physical Examination
Description: Physical examination included assessment of the head, eyes, ears, nose, throat, neck, chest, lungs, abdomen, musculoskeletal, dermatological, cardiovascular/peripheral vascular, and general neurological examination. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for the number of participants with abnormal clinically significant changes in physical examination has been presented.
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Participants | 0

28. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Physical Examination
Description: as for outcome 27
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Participants | 0

29. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected to analyze hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Hematocrit, Hemoglobin, Platelets, and Erythrocytes. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of participants with abnormal clinically significant changes in hematology parameters were reported.
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Participants | 0

30. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Hematology Parameters
Description: as for outcome 29
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Participants | 0

31. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Clinical Chemistry Parameters
Description: Blood samples were collected to analyze clinical chemical parameters: albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, calcium, chloride, creatinine kinase, creatinine, gamma glutamyl transferase, glucose, phosphate, potassium, sodium, total, direct, and indirect bilirubin, protein, urea, and urate. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of Participants with abnormal clinically significant changes in clinical chemistry parameters were reported.
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Participants | 2

32. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Clinical Chemistry Parameters
Description: as for outcome 31
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Participants | 0

33. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Coagulation Parameters
Description: Blood samples were collected to analyze coagulation parameters: activated partial thromboplastin time, prothrombin time international (Intl.) normalized ratio, and prothrombin time. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of Participants with abnormal clinically significant changes in coagulation parameters were reported.
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Participants | 0

34. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Coagulation Parameters
Description: as for outcome 33
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Camlipixant 50 mg + Rabeprazole 20 mg: Participants received a single oral dose of camlipixant 50 mg tablet on Day 1, followed by repeat oral doses of 20 mg rabeprazole enteric-coated tablets, once daily (QD) from Days 4 to 11, with co-administration of a single oral dose of 50 mg camlipixant tablet with rabeprazole enteric-coated tablet on Day 10. There was a washout of at least 3 days between the dose of camlipixant on Day 1 and the dose of rabeprazole on Day 4.was a washout of at least 3 days between the dose of camlipixant on Day 1 and the dose of rifampin on Day 4.
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Participants | 0

35. Secondary Outcome: Part 1: Number of Participants With Abnormal Clinically Significant Changes in Urinalysis
Description: Urine samples were collected to analyze urinalysis parameters: specific gravity and potential of hydrogen (pH). Bilirubin, blood (occult), glucose, ketones, leukocyte esterase, nitrite, protein, urobilinogen were analyzed by dipstick. The dipstick test gives results in a semi-quantitative manner, and results can be read as Negative, Trace, 1+, 2+ indicating proportional concentrations in the urine sample. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of Participants with abnormal clinically significant changes in urinalysis parameters were reported.
Time Frame: Up to Day 13
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Camlipixant 50 mg + Rifampin 600 mg
Number analyzed (Participants) | 16
Participants | 0

36. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinically Significant Changes in Urinalysis
Description: as for outcome 35
Time Frame: Up to Day 12
Population: Safety population consisted of all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Camlipixant 50 mg + Rabeprazole 20 mg
Number analyzed (Participants) | 16
Participants | 0

ADVERSE EVENTS:
Time Frame: Upto Day22 for Part1(Day1 postdose until Day4 predose of rifampin[Camlipixant 50mg];From Day4 dosing until Day11 predose of camlipixant [Rifampin 600mg];From camlipixant dosing on Day11 until end of study[Day22] [Camlipixant 50mg+Rifampin 600mg]. Upto Day21 for Part2(Day1 postdose until Day4 predose of rabeprazole [Camlipixant 50mg];From Day4 dosing until Day10 predose of camlipixant [Rabeprazole 20mg];From camlipixant dosing on Day10 until end of study[Day21] [Camlipixant 50mg+Rabeprazole 20mg]
Description: Safety Population comprised of all participants who received at least one dose of any study drug. Adverse events were reported treatment-wise and part-wise.
Groups:
- Part 1: Camlipixant 50 mg+ Rifampin 600 mg: Participants received repeat oral doses (2*300 mg) of rifampin 600 mg capsules, once daily (QD) from Days 4 to 12, with co-administration of a single oral dose of 50 mg camlipixant tablet with rifampin capsules on Day 11. Participants were followed up for adverse events until end of study (up to Day 22)
Arm/Group | Part 1: Camlipixant 50 mg | Part 1: Rifampin 600 mg | Part 1: Camlipixant 50 mg+ Rifampin 600 mg | Part 2: Camlipixant 50 mg | Part 2 : Rabeprazole 20 mg | Part 2: Camlipixant 50 mg+ Rabeprazole 20 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 14/16 | 2/16 | 4/16 | 3/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Camlipixant 50 mg (N=16) | Part 1: Rifampin 600 mg (N=16) | Part 1: Camlipixant 50 mg+ Rifampin 600 mg (N=16) | Part 2: Camlipixant 50 mg (N=16) | Part 2 : Rabeprazole 20 mg (N=16) | Part 2: Camlipixant 50 mg+ Rabeprazole 20 mg (N=16)
Chromaturia (Renal and urinary disorders) | 0 | 13 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT05899829/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT05899829/SAP_001.pdf